CLINICAL TRIAL: NCT03267992
Title: Observational Study of HGE Health Care Solution COPD Co-Pilot AIR™ Application in Subjects Undergoing the PneumRx® Endobronchial Coil Procedure as Part of EU Registry CLN0014
Brief Title: Chronic Obstructive Pulmonary Disease (COPD) Co-Pilot AIR Substudy of CLN0014
Acronym: Co-Pilot Air
Status: Terminated | Type: Observational
Why Stopped: Study enrollment was prematurely stopped for business reasons.
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: PneumRx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN0020
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: COPD Symptoms After Coil Procedure
Keywords: COPD; Coils; App
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: COPD Co-Pilot AIR App — App. For COPD symptoms after Coil procedure

SUMMARY:
The purpose of undertaking CLN0020, which was a Substudy of the European Coil registry (CLN0014), was to investigate the use of COPD Co-Pilot AIR™, a COPD disease management program manufactured and operated by HGE Health Care Solutions, LLC, in participants undergoing the PneumRx Endobronchial Coil Treatment in a post-market setting.

DETAILED DESCRIPTION:
COPD Co-Pilot AIR™ combines a digital respiratory symptom reporting participant application (an "app") with facilitation of rapid personalized clinical recommendations made by the participant's health care provider and communicated to the participant through the application. COPD Co-Pilot AIR™ provides early identification of an increase in a participant's respiratory symptoms relative to the participant's own baseline symptom profile which in turn enables health care providers to rapidly implement modified treatment plans.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has read, understood, and signed a CLN0020 informed consent form prior to enrollment.
2. Participant is appropriate for Coil treatment per the Conformité Européene (European Conformity [CE])-Mark Approved RePneu Instructions for Use (IFU).
3. Participant has been enrolled in and scheduled for treatment(s) with the PneumRx Endobronchial Coil procedure in the CLN0014 study.
4. Participant's PneumRx Endobronchial Coil procedure is scheduled to occur no fewer than 14 days from enrollment, providing enough time to establish a baseline of their daily symptoms. Ten days minimum of baseline data are required, which is defined as the Run-in period going forward.
5. Participant is willing and able to use a smart phone.

Exclusion Criteria:

1. Participant has undergone a Coil procedure.
2. Participant has had an acute exacerbation of COPD that required hospitalization or emergency room visit or treatment with systemic steroids and/or antibiotics during the 28 days prior to CLN0020 enrollment.
3. Participant has a COPD exacerbation or respiratory illness during the Run-in period that in the judgment of the investigator requires medical intervention (for example, treatment with systemic steroids and/or antibiotics and/or hospitalization).
4. Participant is suffering from terminal illness expected to adversely affect survival in the next 12 months.
5. Participant has a history of non-compliance with medical therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with COPD undergoing the PneumRx Endobronchial Coil Treatment in a post-market setting.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2018-10-20 (Actual)

PRIMARY OUTCOMES:
Rate of COPD Exacerbation | 12 months
  Rate of COPD Exacerbation serious adverse events (SAEs) reported in the 12-month period following the initial Endobronchial Coil procedure for participants enrolled in CLN0020 when compared to CLN0014 participant population that was not managed utilizing COPD Co-Pilot AIR.

SECONDARY OUTCOMES:
Respiratory Related SAEs | 12 months
  Percent of participants experiencing one or more respiratory-related SAEs in the 12-month period following the initial Coil procedure comparing participants enrolled in CLN0020 to non-COPD Co-Pilot AIR participants in CLN0014.
Rate of First Respiratory-Related SAEs | 12 months
  Rate of first respiratory-related SAEs reported in the 12-month period following the initial Coil procedure comparing participants enrolled in CLN0020 to non-COPD Co-Pilot AIR participants enrolled in CLN0014.
Time to First Respiratory-Related SAE | 12 months
  Time to first respiratory-related SAE following the initial Coil procedure comparing participants enrolled in CLN0020 to non-COPD Co-Pilot AIR participants enrolled in CLN0014.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Franzen, MD, Principal Investigator — Klinik für Pneumologie, Zurich
Locations (2):
- Switzerland (2):
  - Hôpitaux Universitaires de Genève (HUG) Service, Geneva
  - UniversitätsSpital, Zurich